CLINICAL TRIAL: NCT05578144
Title: Using "Share Decision Making With Patient Decision Aids" to Help the Infant Family to Decide Whether the Baby Will Receive the Third Primary Dosing Pneumococcal Conjugate Vaccine
Brief Title: Using "SDM With PDAs" to Help Infant Family to Decide the Third Primary Dosing Pneumococcal Conjugate Vaccine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 111HHC-05
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Infants' Family Decide Baby's Vaccine
Keywords: SDM; PDAs; Pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient decision aids group (Experimental): shared decision making with using patient decision aids. (SDM group)
  Interventions: Other: Patients Decision Aids (PDA)
- Control group (No Intervention): oral explanation. (Non-SDM group)

INTERVENTIONS:
Other: Patients Decision Aids (PDA) — Patient Decision Aids (PDA) administer to case group
  Arms: Patient decision aids group

SUMMARY:
Pneumococcal infection is one the common infectious disease in the world. Pneumococcal conjugate vaccine may decrease the incidence of pneumococcal infection. In Taiwan, infants usually received 2 primary dosing pneumococcal conjugate vaccines . The third primary dose of pneumococcal conjugate vaccine is still not included in public health insurance. Some infants in Taiwan did not receive the third primary dose of pneumococcal vaccine. Share decision making (SDM) with patient decision aids (PDA) provide information to infant family and to help them in making decisions about their baby's vaccination. We develop a PDA administered for baby's family to decide whether the baby will receive the third primary dosing pneumococcal conjugate vaccine.

DETAILED DESCRIPTION:
Pneumococcal infection is one of the most major infectious disease that cause morbidity and mortality due to pneumonia, meningitis, acute otitis media, acute rhinosinusitis and septicemia. Although pneumococcal infection may affect people in all ages, children below 5-year-old and adults over 65-year-old are high risk group. Pneumococcal conjugate vaccine has decreased the incidence of pneumococcal infection in the world. Infants usually received 2 primary dosing pneumococcal conjugate vaccines on schedule in Taiwan. The third primary dose of pneumococcal conjugate vaccine is still not included in public health insurance. Many infants' family did not know the information of the third primary dosing pneumococcal conjugate vaccine; and not all of the infants in Taiwan received the third primary dose of pneumococcal vaccine. Share decision making (SDM) with patient decision aids (PDA) is one way to provide information to infants' family and to help them in making decisions about their baby's vaccination. We develop a PDA administered for baby's family to decide whether the baby will receive the third primary dosing pneumococcal conjugate vaccine.

ELIGIBILITY:
Inclusion Criteria:

The 4-month-old baby's family aged between 20 and 80 years old.

Exclusion Criteria:

The baby's family is not suitable; baby's family cannot understand languages what we said; the participants' baby who have fever or contraindication for self-paid third primary PCV.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Decisional conflict | An average of ３month after intervention
  Total scores of decisional conflict scale
Decision-making difficulties | An average of ３month after intervention
  Total scores of decision-making scale

SECONDARY OUTCOMES:
Percentage of the infant's families let baby receiving third primary PCV | An average of ３month after intervention
  vaccination rate

IPD SHARING:
Plan to Share IPD: No